CLINICAL TRIAL: NCT06985888
Title: Clinical Investigation of a New Coating for Urinary Intermittent Catheters in Healthy Volunteers
Brief Title: New Coating for Urinary Intermittent Catheters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CP372
Record Dates: First submitted 2025-04-28; First posted 2025-05-22 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-05

CONDITIONS: Retention, Urinary
MeSH Terms: conditions — Urinary Retention

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Catheterisation with investigational device and Comparator (Other)
  Interventions: Device: SpeediCath® Standard male new coating; Device: SpeediCath® Standard male
- Catheterisation with Comparator and Investigational device (Other)
  Interventions: Device: SpeediCath® Standard male new coating; Device: SpeediCath® Standard male

INTERVENTIONS:
Device: SpeediCath® Standard male new coating — Intermittent catheterization through the urethra draining the bladder, using SpeediCath® Standard male new coating CH12 by HCP
Device: SpeediCath® Standard male — Intermittent catheterization through the urethra draining the bladder, using SpeediCath® Standard male CH 12 by HCP

SUMMARY:
The goal is to confirm, that the newly developed coating is non-inferior to the comparator with respect to the overall discomfort of the catheterisation (assessed by participant).

Participants will attend 3 study site visits and will be catheterised by a HCP at visit 1 and 2 with one of the two catheters in randomisation order. Urine samples will be collected pre- and post catheterisation for assessments.

DETAILED DESCRIPTION:
The primary objective of the study is to confirm that the newly developed investigational coating is non-inferior to the comparator coating with respect to the overall discomfort of catheterisation.

The investigational device is a ready-to-use, sterile, hydrophilic-coated Nelaton male catheter for intermittent catheterisation and based on the standard SpeediCath® male intermittent catheter with a difference in the composition on the coating.

The study is a double-blinded, randomized, crossover study including 32 randomized healthy male volunteers. The total study duration for the individual subject will be between 4-21 days and consists of 3 site visits V0, V1 and V2, and V0 andV1 can be combined

At V1 and V2 the subjects will be catheterized in a hospital setting by a health care professional, with one of the two catheters in a randomized order. Subject will be asked to assess the overall discomfort of the catheterisation on VAS.

ELIGIBILITY:
Inclusion Criteria:

1. Has given written informed consent
2. Is at least 18 years old
3. Has full legal capacity
4. Has self-assessed intact male anatomy with no abnormalities or disease of the lower urinary tract or any surgical procedures performed in the lower urinary tract
5. Is able (assessed by investigator) and willing to adhere to study procedures during study duration.
6. Is able to refrain from using analgesics up to 24 hours prior to catheterisation visits
7. Is negative for haematuria, measured by urine dipstick test of erythrocytes

Exclusion Criteria:

1. Is participating in any other clinical investigation during this investigation, which could affect the results of this investigation, as assessed by investigator.
2. Has previously been randomized in this investigation.
3. Has known hypersensitivity towards any of the devices used in the investigation
4. Is currently experiencing symptoms associated with UTI, as assessed by investigator.
5. Has known impaired sensation of the urethra

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2025-05-06 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Overall discomfort of the catheterisation | immediately after the procedure
  assessed by subject using VAS

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, Rigshospitalet, Copenhagen, Denmark